CLINICAL TRIAL: NCT06302894
Title: The Effect of Nursing Intervention Program for Problematic Internet User Adolescents on Appropriate Internet Use, Loneliness and Family Cohesion
Brief Title: The Effect of the Nursing Intervention Program on Adolescent Problematic Internet Users
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Eda Çeker, lecturer, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BAIBU-SBF-EC-01
Record Dates: First submitted 2024-03-01; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Internet Addiction Disorder
Keywords: Family Cohesion Scale; Internet Addiction Scale; Loneliness Scale for Children
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Internet addiction scale, family harmony scale and loneliness scale for children will be applied to the control group after 6 weeks without any intervention.
- Experimental group (Experimental): In order to reduce problematic internet use and protect the experimental group from addiction, different online applications and trainings based on the Health Belief Model, enriched with web 2.0 technologies, will be provided and followed every week (6 weeks in total).
  At the end of 6 weeks, the internet addiction scale, family harmony scale and loneliness scale for children will be administered.
  Interventions: Behavioral: Self-sufficiency

INTERVENTIONS:
Behavioral: Self-sufficiency — Rewarding positive behavior and developing alternative behaviors towards obstacles such as feeling restless, depressed or angry if internet use is reduced or controlled.
  Arms: Experimental group

SUMMARY:
In this study; The effect of the nursing intervention program (education enriched with web 2.0 tools based on the Health Belief Model) on problematic internet use, loneliness and family harmony in adolescents who use the internet with problems will be determined.

DETAILED DESCRIPTION:
In this study; The effect of the nursing intervention program (education enriched with web 2.0 tools based on the Health Belief Model) on problematic internet use, loneliness and family harmony in adolescents who use the internet with problems will be determined. This research is a cross-sectional randomized controlled experimental study with a cross-sectional type in the first stage and a pretest-posttest in the second stage.

ELIGIBILITY:
Inclusion Criteria:

1. Being a secondary school student,
2. Agreeing to participate in the research,
3. Being open to communication and cooperation,
4. Can use web 2.0 tools via smartphone or computer

Exclusion Criteria:

- Having a score of less than 50 points and above 79 points on the Internet addiction scale.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Internet Addiction Scale | 5 weeks
  In the first stage, pre-measurement will be applied to all students in the sample. In the first stage, students who score between 50-79 (risky internet use behavior / limited symptoms) on the Internet Addiction Scale of secondary school students will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Eda Ceker, Lecturer, Principal Investigator — Bolu Abant İzzet Baysal University Faculty of Health Sciences
Locations (1):
- Bolu Abant İzzet Baysal University Faculty of Health Sciences, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No